CLINICAL TRIAL: NCT05696080
Title: A Phase 3, Randomized, Double-blind, Active Comparator-controlled Clinical Study to Evaluate the Safety, Tolerability, and Immunogenicity of V116 in Pneumococcal Vaccine-naïve Adults 18 to 64 Years of Age With Increased Risk for Pneumococcal Disease.
Brief Title: Safety and Immunogenicity of V116 in Adults With Increased Risk for Pneumococcal Disease (V116-008)
Acronym: STRIDE-8
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V116-008; V116-008 (Other: MSD); jRCT2061220106 (Registry Identifier: jRCT); 2022-502791-22 (Other: EU CT); U1111-1282- 1460 (Other: UTN)
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Results first posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Pneumococcal Infection
MeSH Terms: conditions — Pneumococcal Infections | interventions — 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- V116 + Placebo (Experimental): Participants administered a single intramuscular (IM) dose of V116 on Day 1, and single IM dose of placebo on Week 8.
  Interventions: Biological: V116; Biological: Placebo
- PCV15 + PPSV23 (Active Comparator): Participants administered a single IM dose of PCV15 on Day 1, and a single IM dose of PPSV23 on Week 8.
  Interventions: Biological: PCV15; Biological: PPSV23

INTERVENTIONS:
Biological: V116 — Pneumococcal 21-valent conjugate vaccine with 4 μg of each of the following pneumococcal polysaccharides (PnPs) antigen: 3, 6A, 7F, 8, 9N, 10A, 11A, 12F, 15A, 15C, 16F, 17F, 19A, 20, 22F, 23A, 23B, 24F, 31, 33F, and 35B in each 0.5 mL sterile solution
  Other Names: Pneumococcal 21-valent Conjugate Vaccine
  Arms: V116 + Placebo
Biological: Placebo — Saline in each 0.5 mL sterile solution
  Arms: V116 + Placebo
Biological: PCV15 — Pneumococcal 15-valent conjugate vaccine with 2 μg of each of the following PnPs antigen: 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F; and 4 μg of PnPs antigen 6B in each 0.5 mL sterile suspension
  Other Names: VAXNEUVANCE™
  Arms: PCV15 + PPSV23
Biological: PPSV23 — Pneumococcal 23-valent polyvalent vaccine with 25 μg of each of the following PnPs antigen: 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F, and 33F in each 0.5 mL sterile solution
  Other Names: PNEUMOVAX™23
  Arms: PCV15 + PPSV23

SUMMARY:
The primary objectives of this study are to evaluate the safety and tolerability of the pneumococcal 21 valent conjugate vaccine (V116), and to evaluate the serotype-specific opsonophagocytic activity (OPA) post-vaccination with V116 and PCV15 (a pneumococcal conjugate vaccine that includes 15 serotypes) + PPSV23 (comprised of the polysaccharides from 23 of the serotypes causing disease in adults) post-vaccination within each vaccination group separately.

ELIGIBILITY:
Inclusion Criteria:

* Has documented result(s) of ≥1 of the following risk conditions for pneumococcal disease: diabetes mellitus, receiving treatment with ≥1 approved antidiabetic medication, with all Hemoglobin A1c (HbA1c) measurements ≤9% within 6 months before first study vaccination; compensated chronic liver disease; diagnosis of chronic obstructive pulmonary disease (COPD) managed per local guidelines; diagnosis of mild or moderate persistent asthma managed per local guidelines; confirmed diagnosis of chronic heart disease managed per local guidelines; confirmed diagnosis of chronic kidney disease (>3 months duration).
* Is receiving stable medical management for the listed risk conditions for ≥3 months with no anticipated major change in treatment expected for the duration of the study and with ≤1 hospitalization directly related to the risk condition.
* Female Is not a participant of childbearing potential (POCBP); or if a POCBP Uses an acceptable contraceptive method or is abstinent from penile-vaginal intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis); their medical history, menstrual history, and recent sexual activity has been reviewed by the investigator.

Exclusion Criteria:

* Has a history of active hepatitis.
* Has a history of diabetic ketoacidosis or 2 or more episodes of severe, symptomatic hypoglycemia within 3 months before first study vaccination (Day 1).
* Has a history of myocardial infarction, acute coronary syndrome, transient ischemic attack, or ischemic or hemorrhagic stroke within 3 months before first study vaccination (Day 1).
* Has a history of severe pulmonary hypertension with World Health Organization (WHO) functional class ≥3 or history of Eisenmenger syndrome
* Has a history of autoimmune related chronic kidney disease, chronic kidney failure, a reversible cause of kidney disease, nephrotic syndrome, or any ineligible Kidney Disease: Improving Global Outcomes (KDIGO)-recommended stage of glomerular filtration rate (GFR) and Albuminuria
* Has a history of invasive pneumococcal disease (IPD) (positive blood culture, positive cerebrospinal fluid culture, or positive culture at another sterile site) or known history of other culture-positive pneumococcal disease within 3 years before first study vaccination (Day 1).
* Has a known hypersensitivity to any component of V116, PCV15, or PPSV23, including diphtheria toxoid.
* Has a known or suspected impairment of immunological function including, but not limited to, congenital or acquired immunodeficiency, documented human immunodeficiency virus (HIV) infection, functional or anatomic asplenia, or autoimmune disease.
* Has a coagulation disorder contraindicating intramuscular (IM) vaccination.
* Had a recent febrile illness or received antibiotic therapy for any acute illness occurring within 72 hours before receipt of any study vaccine.
* Has a known malignancy that is progressing or has required active treatment <3 years before randomization.
* Has planned organ transplantation (heart, liver, lung, kidney, or pancreas) or other planned major surgical procedure during the duration of this study.
* Has expected survival for <1 year.
* Has received any prior pneumococcal vaccine or is expected to receive any pneumococcal vaccine during the study outside the protocol.
* Has received systemic corticosteroids (prednisone equivalent of ≥20 mg/day) for ≥14 consecutive days and has not completed intervention ≥14 days before receipt of study vaccine at Visit 2 (Day 1).
* Is currently receiving systemic immunosuppressive therapy, including chemotherapeutic agents or other immunotherapies/immunomodulators used to treat cancer or other conditions, and interventions associated with organ or bone marrow transplantation, or autoimmune disease.
* Has received any non-live vaccine ≤14 days before receipt of any study vaccine or is scheduled to receive any non-live vaccine ≤30 days after receipt of any study vaccine.
* Has received any live virus vaccine (including severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) live virus vaccines) ≤30 days before receipt of any study vaccine or is scheduled to receive any live virus vaccine ≤30 days after receipt of any study vaccine
* Has received a blood transfusion or blood products, including immunoglobulin ≤6 months before receipt of any study vaccine or is scheduled to receive a blood transfusion or blood product ≤30 days after receipt of any study vaccine.
* Is receiving chronic home oxygen therapy.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 518 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director, Study Director — Merck Sharp & Dohme LLC
Locations (44):
- United States (8):
  - Aventiv Research ( Site 0022), Mesa, Arizona
  - Indago Research & Health Center, Inc ( Site 0002), Hialeah, Florida
  - Triple O Research Institute, P.A ( Site 0011), West Palm Beach, Florida
  - SKY Integrative Medical Center/SKYCRNG ( Site 0012), Ridgeland, Mississippi
  - Mid Hudson Medical Research ( Site 0008), New Windsor, New York
  - Holston Medical Group ( Site 0010), Kingsport, Tennessee
  - EmVenio Research ( Site 0018), Fort Worth, Texas
  - Wenatchee Valley Hospital ( Site 0019), Wenatchee, Washington
- Australia (2):
  - Holdsworth House Medical Practice ( Site 0402), Darlinghurst, New South Wales
  - Royal Brisbane and Women's Hospital ( Site 0400), Brisbane, Queensland
- Canada (7):
  - G A Research Associates ( Site 0100), Moncton, New Brunswick
  - Hamilton Medical Research Group ( Site 0107), Hamilton, Ontario
  - Milestone Research Inc. ( Site 0106), London, Ontario
  - Manna Research Mirabel ( Site 0105), Mirabel, Quebec
  - Clinique de médecine Urbaine du Quartier Latin ( Site 0111), Montreal, Quebec
  - Diex Recherche Trois-Rivieres ( Site 0110), Trois-Rivières, Quebec
  - Diex Recherche Victoriavile Inc. ( Site 0102), Victoriaville, Quebec
- Chile (7):
  - Centro de Investigación del Maule-Centro de Investigación 2 ( Site 1010), Talca, Maule Region
  - Universidad San Sebastian - Providencia ( Site 1003), Providencia, Region M. de Santiago
  - Centro de Investigaciones Medicas Respiratorias (CIMER) ( Site 1008), Santiago, Region M. de Santiago
  - Centro de Investigacion Clinicadela Universidad Catolica ( Site 1004), Santiago, Region M. de Santiago
  - Universidad de Chile - Hospital Clínico Universidad de Chile-Cardiology ( Site 1006), Santiago, Region M. de Santiago
  - CESFAM Esmeralda ( Site 1009), Santiago, Region M. de Santiago
  - Hospital Dr. Hernán Henríquez Aravena ( Site 1001), Temuco, Región de la Araucanía
- Japan (2):
  - Medical corporation Applied Bio-Pharmatech Kurume Clinical Pharmacology Clinic ( Site 0200), Kurume, Fukuoka
  - Shimonoseki Medical Center ( Site 0201), Shimonoseki, Yamaguchi
- New Zealand (6):
  - Pacific Clinical Research Network - Rotorua ( Site 0500), Rotorua, Bay of Plenty
  - P3 Research - Tauranga ( Site 0507), Tauranga, Bay of Plenty
  - CGM Research Trust ( Site 0505), Christchurch, Canterbury
  - Pacific Clinical Research Network - Forte ( Site 0501), Christchurch, Canterbury
  - P3 Research - Lower Hutt ( Site 0508), Lower Hutt, Wellington Region
  - P3 Research - Wellington ( Site 0503), Wellington
- Poland (7):
  - IN VIVO ( Site 0601), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Centrum Medyczne Pratia Bydgoszcz-Centrum Medyczne Pratia Bydgoszcz ( Site 0607), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - MICS Centrum Medyczne Torun ( Site 0606), Torun, Kuyavian-Pomeranian Voivodeship
  - Centrum Medyczne Medyk ( Site 0602), Rzeszów, Podkarpackie Voivodeship
  - Centrum Medyczne Pratia Katowice ( Site 0604), Katowice, Silesian Voivodeship
  - Clinical Medical Research ( Site 0605), Katowice, Silesian Voivodeship
  - Clinmedica Research Sp. z. o. o. ( Site 0603), Skierniewice, Łódź Voivodeship
- South Korea (5):
  - Hallym University Sacred Heart Hospital ( Site 0303), Anyang-si, Kyonggi-do
  - Korea University Anam Hospital ( Site 0305), Seoul
  - Seoul National University Hospital ( Site 0300), Seoul
  - Konkuk University Medical Center ( Site 0302), Seoul
  - Hallym University Kangdong Sacred Heart Hospital ( Site 0301), Seoul

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26329&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pneumococcal vaccine-naïve adults 18 to 64 years of age (inclusive) with increased risk of pneumococcal disease were enrolled in this study. Participants must have had documented results of ≥ 1 of the following risk conditions: diabetes mellitus, chronic heart disease, chronic kidney disease, chronic liver disease, and/or chronic lung disease. Participants with comorbidities were eligible if the conditions were assessed to be stable as per the investigator's judgment.
Groups:
- V116 + Placebo: Pneumococcal vaccine-naïve adult participants (18-64 years of age) received a 0.5mL single intramuscular (IM) dose of pneumococcal 21-valent conjugate vaccine (V116) at Visit 2 (Day 1) and a 0.5mL single IM dose of Placebo (sterile saline) at Visit 5 (Week 8).
- PCV15 + PPSV23: Pneumococcal vaccine-naïve adult participants (18-64 years of age) received a 0.5mL single IM dose of a pneumococcal 15-valent conjugate vaccine (PCV15) at Visit 2 (Day 1) and a 0.5mL single IM dose of pneumococcal vaccine comprised of polysaccharides from 23 of the serotypes causing disease in adults (PPSV23) at Visit 5 (Week 8).
Period: Overall Study
Arm/Group | V116 + Placebo | PCV15 + PPSV23
Started | 387 | 131
Vaccinated With V116 at Visit 2 | 386 | 0
Vaccinated With PCV15 at Visit 2 | 0 | 130
Vaccinated With Placebo at Visit 5 | 374 | 0
Vaccinated With PPSV23 at Visit 5 | 0 | 128
Completed | 372 | 129
Not Completed | 15 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Randomized By Mistake Without Study Treatment | 0 | 1
Not completed — Withdrawal by Subject | 12 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V116 + Placebo | PCV15 + PPSV23 | Total
Number analyzed (Participants) | 387 | 131 | 518
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.4 (9.6) | 53.3 (8.9) | 52.6 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178 | 55 | 233
  Male | 209 | 76 | 285
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 101 | 35 | 136
  Not Hispanic or Latino | 281 | 94 | 375
  Unknown or Not Reported | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 58 | 18 | 76
  Native Hawaiian or Other Pacific Islander | 10 | 8 | 18
  Black or African American | 16 | 2 | 18
  White | 294 | 101 | 395
  More than one race | 8 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Solicited Injection-site Adverse Events (AEs) From Day 1 Through Day 5 Post-vaccination
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants with solicited injection-site AEs was assessed following any vaccination. Solicited injection-site AEs consist of the following: pain/tenderness, redness/erythema, and swelling.
Time Frame: Up to 5 days following each vaccination
Population: All participants who were randomized and received at least 1 dose of study intervention. Participants were included in the intervention group according to the study intervention actually received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V116 + Placebo | PCV15 + PPSV23
Number analyzed (Participants) | 386 | 130
Percentage of participants
  Injection site erythema | 9.1 [6.4 to 12.4] | 25.4 [18.2 to 33.8]
  Injection site pain | 51.8 [46.7 to 56.9] | 78.5 [70.4 to 85.2]
  Injection site swelling | 8.0 [5.5 to 11.2] | 35.4 [27.2 to 44.2]

2. Primary Outcome: Participants With Solicited Systemic AEs From Day 1 Through Day 5 Post-vaccination
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants with solicited systemic AEs was assessed following any vaccination. Solicited systemic AEs consist of the following: fatigue (tiredness), headache, myalgia (muscle aches), and pyrexia (maximum temperature >= 100.4 °F/38.0 °C).
Time Frame: Up to 5 days following each vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V116 + Placebo | PCV15 + PPSV23
Number analyzed (Participants) | 386 | 130
Percentage of participants
  Fatigue | 30.3 [25.8 to 35.2] | 45.4 [36.6 to 54.3]
  Headache | 22.3 [18.2 to 26.8] | 26.2 [18.8 to 34.6]
  Myalgia | 10.9 [8.0 to 14.4] | 15.4 [9.7 to 22.8]
  Pyrexia | 3.1 [1.6 to 5.4] | 4.6 [1.7 to 9.8]

3. Primary Outcome: Participants With Vaccine-related Serious Adverse Events (SAEs) From Day 1 Through The Duration of Participation in The Study
Description: A vaccine-related SAE is any untoward medical consequence that results in death, is life-threatening, requires inpatient hospitalization or prolongs existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is another important medical event, which is determined by the investigator to be related to the vaccine. The percentage of participants with SAEs was assessed following any vaccination.
Time Frame: Up to 194 days following Visit 2 (Day 1)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V116 + Placebo | PCV15 + PPSV23
Number analyzed (Participants) | 386 | 130
Percentage of participants | 0.0 [0.0 to 1.0] | 0.0 [0.0 to 2.8]

4. Primary Outcome: Serotype-specific Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) for Pneumococcal Serotypes Contained in V116
Description: The serotype specific OPA GMTs for the pneumococcal serotypes were determined using the multiplex opsonophagocytic assay (MOPA). The point estimate was calculated by exponentiating the estimates of the mean of the natural log values and within-group 95% CIs were obtained by exponentiating the CIs of the mean of the natural log values based on the t-distribution. The 13 common pneumococcal serotypes in both V116 and PCV15 + PPSV23 were as follows: 3, 6A, 7F, 8, 9N, 10A, 11A, 12F, 17F, 19A, 20A, 22F, and 33F. The 8 unique pneumococcal serotypes in V116 were as follows: 15A, 15C, 16F, 23A, 23B, 24F, 31, and 35B.
Time Frame: 30 days following V116 [Day 30] for the V116 + Placebo group and 30 days following PPSV23 [Week 12] for the PCV15 + PPSV23 group.
Population: The population analyzed was all randomized participants without deviations from the protocol that may substantially affect the results of the immunogenicity endpoints. Deviations include but are not limited to the following: failure to receive the study vaccine, receiving incorrect clinical material per the randomization schedule, or taking prohibited medications or vaccines prior to vaccination or blood sample collection outside the designated window.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | V116 + Placebo | PCV15 + PPSV23
Number analyzed (Participants) | 386 | 130
Titers
  Serotype 3: number analyzed (Participants) | 352 | 104
  Serotype 3 | 216.2 [188.6 to 247.8] | 192.9 [156.7 to 237.4]
  Serotype 6A: number analyzed (Participants) | 347 | 92
  Serotype 6A | 3734.9 [3204.3 to 4353.4] | 2443.8 [1779.0 to 3357.1]
  Serotype 7F: number analyzed (Participants) | 355 | 109
  Serotype 7F | 4261.2 [3781.6 to 4801.6] | 3218.5 [2627.3 to 3942.6]
  Serotype 8: number analyzed (Participants) | 357 | 106
  Serotype 8 | 3460.8 [3083.1 to 3884.7] | 3406.4 [2635.8 to 4402.2]
  Serotype 9N: number analyzed (Participants) | 354 | 107
  Serotype 9N | 7553.9 [6664.1 to 8562.5] | 4548.4 [3696.8 to 5596.2]
  Serotype 10A: number analyzed (Participants) | 355 | 107
  Serotype 10A | 4502.0 [3933.7 to 5152.4] | 2542.0 [1897.0 to 3406.2]
  Serotype 11A: number analyzed (Participants) | 358 | 106
  Serotype 11A | 3761.7 [3375.8 to 4191.7] | 1697.2 [1338.4 to 2152.2]
  Serotype 12F: number analyzed (Participants) | 356 | 107
  Serotype 12F | 2432.3 [2082.7 to 2840.6] | 1364.5 [956.1 to 1947.4]
  Serotype 17F: number analyzed (Participants) | 354 | 104
  Serotype 17F | 10425.3 [9099.2 to 11944.7] | 4331.7 [3248.3 to 5776.3]
  Serotype 19A: number analyzed (Participants) | 356 | 106
  Serotype 19A | 2837.2 [2535.2 to 3175.2] | 2437.2 [2008.5 to 2957.5]
  Serotype 20A: number analyzed (Participants) | 357 | 99
  Serotype 20A | 8091.5 [7169.4 to 9132.3] | 3749.8 [2932.4 to 4795.2]
  Serotype 22F: number analyzed (Participants) | 357 | 108
  Serotype 22F | 4432.7 [3914.2 to 5020.0] | 2717.4 [2201.7 to 3353.8]
  Serotype 33F: number analyzed (Participants) | 347 | 101
  Serotype 33F | 24512.8 [21149.8 to 28410.7] | 11395.1 [8884.5 to 14615.3]
  Serotype 15A: number analyzed (Participants) | 353 | 104
  Serotype 15A | 7274.6 [6398.7 to 8270.4] | 1791.8 [1361.7 to 2357.8]
  Serotype 15C: number analyzed (Participants) | 353 | 107
  Serotype 15C | 7923.1 [6726.7 to 9332.3] | 2269.8 [1651.8 to 3118.9]
  Serotype 16F: number analyzed (Participants) | 356 | 105
  Serotype 16F | 9546.6 [8396.2 to 10854.6] | 1626.2 [1224.4 to 2159.8]
  Serotype 23A: number analyzed (Participants) | 346 | 100
  Serotype 23A | 5875.3 [5005.5 to 6896.2] | 1493.9 [1009.1 to 2211.5]
  Serotype 23B: number analyzed (Participants) | 354 | 108
  Serotype 23B | 2316.9 [1925.9 to 2787.3] | 117.0 [73.4 to 186.4]
  Serotype 24F: number analyzed (Participants) | 354 | 92
  Serotype 24F | 5677.1 [5098.2 to 6321.8] | 1666.8 [1257.6 to 2209.1]
  Serotype 31: number analyzed (Participants) | 359 | 105
  Serotype 31 | 5803.9 [4991.8 to 6748.1] | 360.7 [233.0 to 558.5]
  Serotype 35B: number analyzed (Participants) | 347 | 104
  Serotype 35B | 13141.3 [11584.8 to 14906.9] | 1812.1 [1408.6 to 2331.2]

5. Secondary Outcome: Serotype-specific Immunoglobulin G (IgG) Geometric Mean Concentrations (GMCs) for Pneumococcal Serotypes Contained in V116
Description: The serotype specific IgG GMCs for the pneumococcal serotypes were determined using pneumococcal electrochemiluminescence assay (PnECL). The point estimate was calculated by exponentiating the estimates of the mean of the natural log values and within-group 95% CIs were obtained by exponentiating the CIs of the mean of the natural log values based on the t-distribution. The 13 common pneumococcal serotypes in both V116 and PCV15 + PPSV23 were as follows: 3, 6A, 7F, 8, 9N, 10A, 11A, 12F, 17F, 19A, 20A, 22F, and 33F. The 8 unique pneumococcal serotypes in V116 were as follows: 15A, 15C, 16F, 23A, 23B, 24F, 31, and 35B.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V116 + Placebo | PCV15 + PPSV23
Number analyzed (Participants) | 386 | 130
μg/mL
  Serotype 3: number analyzed (Participants) | 366 | 112
  Serotype 3 | 0.77 [0.69 to 0.87] | 0.79 [0.68 to 0.92]
  Serotype 6A: number analyzed (Participants) | 367 | 112
  Serotype 6A | 4.57 [3.82 to 5.48] | 5.83 [4.23 to 8.03]
  Serotype 7F: number analyzed (Participants) | 367 | 112
  Serotype 7F | 8.77 [7.65 to 10.06] | 6.95 [5.39 to 8.96]
  Serotype 8: number analyzed (Participants) | 367 | 112
  Serotype 8 | 10.20 [8.89 to 11.71] | 12.50 [9.68 to 16.14]
  Serotype 9N: number analyzed (Participants) | 367 | 112
  Serotype 9N | 7.53 [6.42 to 8.83] | 4.35 [3.35 to 5.66]
  Serotype 10A: number analyzed (Participants) | 367 | 112
  Serotype 10A | 12.18 [10.36 to 14.32] | 6.88 [5.07 to 9.34]
  Serotype 11A: number analyzed (Participants) | 367 | 112
  Serotype 11A | 7.78 [6.80 to 8.89] | 4.04 [3.22 to 5.07]
  Serotype 12F: number analyzed (Participants) | 367 | 112
  Serotype 12F | 1.90 [1.58 to 2.28] | 0.84 [0.60 to 1.18]
  Serotype 17F: number analyzed (Participants) | 367 | 112
  Serotype 17F | 17.35 [15.06 to 19.98] | 8.20 [6.32 to 10.64]
  Serotype 19A: number analyzed (Participants) | 367 | 112
  Serotype 19A | 9.11 [7.98 to 10.41] | 10.88 [8.70 to 13.60]
  Serotype 20A: number analyzed (Participants) | 367 | 112
  Serotype 20A | 19.51 [16.73 to 22.75] | 13.38 [10.27 to 17.43]
  Serotype 22F: number analyzed (Participants) | 367 | 112
  Serotype 22F | 5.17 [4.44 to 6.02] | 3.98 [3.08 to 5.14]
  Serotype 33F: number analyzed (Participants) | 367 | 112
  Serotype 33F | 15.38 [13.23 to 17.88] | 11.40 [8.99 to 14.46]
  Serotype 15A: number analyzed (Participants) | 367 | 112
  Serotype 15A | 14.65 [12.52 to 17.13] | 2.37 [1.77 to 3.18]
  Serotype 15C: number analyzed (Participants) | 367 | 112
  Serotype 15C | 14.48 [12.07 to 17.38] | 5.42 [3.98 to 7.37]
  Serotype 16F: number analyzed (Participants) | 367 | 111
  Serotype 16F | 2.90 [2.48 to 3.38] | 0.27 [0.21 to 0.35]
  Serotype 23A: number analyzed (Participants) | 367 | 112
  Serotype 23A | 3.85 [3.18 to 4.66] | 0.79 [0.56 to 1.11]
  Serotype 23B: number analyzed (Participants) | 367 | 112
  Serotype 23B | 6.62 [5.75 to 7.63] | 1.46 [1.09 to 1.96]
  Serotype 24F: number analyzed (Participants) | 367 | 112
  Serotype 24F | 5.18 [4.17 to 6.43] | 0.34 [0.26 to 0.43]
  Serotype 31: number analyzed (Participants) | 367 | 112
  Serotype 31 | 3.27 [2.83 to 3.79] | 0.38 [0.29 to 0.49]
  Serotype 35B: number analyzed (Participants) | 367 | 112
  Serotype 35B | 19.78 [17.38 to 22.50] | 1.55 [1.27 to 1.90]

6. Secondary Outcome: Serotype-specific Geometric Mean Fold Rises (GMFRs) for OPA Responses From Baseline to Post-vaccination With V116 and PCV15 + PPSV23
Description: The geometric mean fold rise (GMFR) from baseline to post-vaccination in serotype specific OPA GMTs was determined using MOPA. The within-group 95% confidence intervals (Cis) were obtained by exponentiating the CIs of the mean of the natural log values based on the t-distribution. The 13 common pneumococcal serotypes in both V116 and PCV15 + PPSV23 were as follows: 3, 6A, 7F, 8, 9N, 10A, 11A, 12F, 17F, 19A, 20A, 22F, and 33F. The 8 unique pneumococcal serotypes in V116 were as follows: 15A, 15C, 16F, 23A, 23B, 24F, 31, and 35B.
Time Frame: Baseline (Day 1) and postvaccination (30 days following V116 [Day 30] for the V116 + Placebo group and 30 days following PPSV23 [Week 12] for the PCV15 + PPSV23 group)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V116 + Placebo | PCV15 + PPSV23
Number analyzed (Participants) | 386 | 130
Ratio
  Serotype 3: number analyzed (Participants) | 334 | 102
  Serotype 3 | 8.3 [7.2 to 9.5] | 6.1 [4.8 to 7.7]
  Serotype 6A: number analyzed (Participants) | 297 | 82
  Serotype 6A | 22.8 [18.6 to 28.0] | 17.1 [11.9 to 24.7]
  Serotype 7F: number analyzed (Participants) | 341 | 107
  Serotype 7F | 20.4 [16.9 to 24.6] | 10.5 [7.5 to 14.7]
  Serotype 8: number analyzed (Participants) | 344 | 103
  Serotype 8 | 25.7 [21.1 to 31.2] | 25.2 [17.0 to 37.1]
  Serotype 9N: number analyzed (Participants) | 336 | 107
  Serotype 9N | 12.6 [10.6 to 15.0] | 7.2 [5.5 to 9.5]
  Serotype 10A: number analyzed (Participants) | 327 | 98
  Serotype 10A | 19.9 [16.1 to 24.5] | 10.7 [7.2 to 15.8]
  Serotype 11A: number analyzed (Participants) | 326 | 100
  Serotype 11A | 20.7 [16.6 to 25.8] | 6.8 [4.6 to 10.1]
  Serotype 12F: number analyzed (Participants) | 343 | 107
  Serotype 12F | 95.0 [79.9 to 113.0] | 48.6 [32.5 to 72.6]
  Serotype 17F: number analyzed (Participants) | 327 | 101
  Serotype 17F | 28.4 [23.6 to 34.2] | 13.1 [9.5 to 18.1]
  Serotype 19A: number analyzed (Participants) | 337 | 102
  Serotype 19A | 9.7 [8.2 to 11.5] | 9.9 [7.2 to 13.6]
  Serotype 20A: number analyzed (Participants) | 335 | 97
  Serotype 20A | 8.5 [7.2 to 10.0] | 3.8 [3.0 to 5.0]
  Serotype 22F: number analyzed (Participants) | 322 | 102
  Serotype 22F | 15.1 [12.2 to 18.7] | 9.1 [6.0 to 13.7]
  Serotype 33F: number analyzed (Participants) | 330 | 100
  Serotype 33F | 12.3 [10.4 to 14.5] | 5.5 [4.1 to 7.2]
  Serotype 15A: number analyzed (Participants) | 309 | 95
  Serotype 15A | 10.4 [8.6 to 12.5] | 2.4 [1.8 to 3.2]
  Serotype 15C: number analyzed (Participants) | 335 | 105
  Serotype 15C | 52.8 [42.1 to 66.2] | 18.3 [12.2 to 27.4]
  Serotype 16F: number analyzed (Participants) | 334 | 96
  Serotype 16F | 8.6 [7.3 to 10.1] | 1.6 [1.2 to 2.0]
  Serotype 23A: number analyzed (Participants) | 261 | 76
  Serotype 23A | 14.5 [11.4 to 18.6] | 4.3 [2.7 to 6.8]
  Serotype 23B: number analyzed (Participants) | 341 | 106
  Serotype 23B | 83.6 [66.4 to 105.3] | 6.2 [4.3 to 9.0]
  Serotype 24F: number analyzed (Participants) | 293 | 81
  Serotype 24F | 4.0 [3.4 to 4.7] | 0.9 [0.7 to 1.2]
  Serotype 31: number analyzed (Participants) | 344 | 99
  Serotype 31 | 23.2 [18.4 to 29.1] | 1.5 [1.2 to 2.0]
  Serotype 35B: number analyzed (Participants) | 337 | 102
  Serotype 35B | 7.2 [6.3 to 8.3] | 1.2 [1.0 to 1.4]

7. Secondary Outcome: Serotype-specific GMFRs for IgG Responses From Baseline to Post-vaccination With V116 and PCV15 + PPSV23
Description: The GMFR from baseline to post-vaccination in serotype specific IgG GMCs was determined using Pn electrochemiluminescence (ECL) assay. The within-group 95% confidence intervals (Cis) were obtained by exponentiating the CIs of the mean of the natural log values based on the t-distribution. The 13 common pneumococcal serotypes in both V116 and PCV15 + PPSV23 were as follows: 3, 6A, 7F, 8, 9N, 10A, 11A, 12F, 17F, 19A, 20A, 22F, and 33F. The 8 unique pneumococcal serotypes in V116 were as follows: 15A, 15C, 16F, 23A, 23B, 24F, 31, and 35B.
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V116 + Placebo | PCV15 + PPSV23
Number analyzed (Participants) | 386 | 130
Ratio
  Serotype 3: number analyzed (Participants) | 365 | 111
  Serotype 3 | 5.2 [4.7 to 5.8] | 4.5 [3.8 to 5.4]
  Serotype 6A: number analyzed (Participants) | 366 | 111
  Serotype 6A | 16.2 [13.9 to 18.9] | 20.1 [15.5 to 26.0]
  Serotype 7F: number analyzed (Participants) | 366 | 111
  Serotype 7F | 19.0 [16.8 to 21.5] | 12.8 [10.2 to 16.2]
  Serotype 8: number analyzed (Participants) | 366 | 111
  Serotype 8 | 14.8 [12.9 to 17.0] | 15.5 [11.5 to 21.0]
  Serotype 9N: number analyzed (Participants) | 366 | 111
  Serotype 9N | 19.2 [16.8 to 22.0] | 9.9 [7.9 to 12.5]
  Serotype 10A: number analyzed (Participants) | 366 | 111
  Serotype 10A | 20.1 [17.6 to 23.0] | 11.0 [8.6 to 13.9]
  Serotype 11A: number analyzed (Participants) | 366 | 111
  Serotype 11A | 11.7 [10.3 to 13.3] | 5.6 [4.5 to 7.0]
  Serotype 12F: number analyzed (Participants) | 366 | 111
  Serotype 12F | 17.7 [15.3 to 20.5] | 8.1 [6.2 to 10.6]
  Serotype 17F: number analyzed (Participants) | 366 | 111
  Serotype 17F | 29.6 [25.9 to 33.8] | 13.9 [10.9 to 17.6]
  Serotype 19A: number analyzed (Participants) | 366 | 111
  Serotype 19A | 7.1 [6.3 to 8.0] | 8.1 [6.5 to 10.0]
  Serotype 20A: number analyzed (Participants) | 366 | 111
  Serotype 20A | 15.1 [13.2 to 17.2] | 8.7 [7.0 to 10.8]
  Serotype 22F: number analyzed (Participants) | 366 | 111
  Serotype 22F | 19.7 [17.0 to 22.8] | 13.2 [10.2 to 17.3]
  Serotype 33F: number analyzed (Participants) | 366 | 111
  Serotype 33F | 14.7 [13.0 to 16.6] | 11.0 [8.8 to 13.8]
  Serotype 15A: number analyzed (Participants) | 366 | 111
  Serotype 15A | 23.6 [20.6 to 27.1] | 3.7 [3.0 to 4.6]
  Serotype 15C: number analyzed (Participants) | 366 | 110
  Serotype 15C | 24.2 [20.8 to 28.2] | 9.2 [7.3 to 11.7]
  Serotype 16F: number analyzed (Participants) | 366 | 110
  Serotype 16F | 16.0 [14.1 to 18.1] | 1.6 [1.4 to 1.9]
  Serotype 23A: number analyzed (Participants) | 366 | 111
  Serotype 23A | 20.9 [18.2 to 24.0] | 3.8 [2.9 to 4.9]
  Serotype 23B: number analyzed (Participants) | 366 | 111
  Serotype 23B | 16.6 [14.3 to 19.2] | 3.7 [3.0 to 4.6]
  Serotype 24F: number analyzed (Participants) | 366 | 111
  Serotype 24F | 18.0 [15.5 to 20.9] | 1.1 [1.1 to 1.2]
  Serotype 31: number analyzed (Participants) | 366 | 111
  Serotype 31 | 14.4 [12.7 to 16.4] | 1.5 [1.4 to 1.7]
  Serotype 35B: number analyzed (Participants) | 366 | 111
  Serotype 35B | 12.8 [11.3 to 14.5] | 1.0 [1.0 to 1.1]

8. Secondary Outcome: Percentage of Participants With ≥4-fold Change From Baseline to Post-vaccination With V116 and PCV15 + PPSV23 in Serotype Specific OPA Responses for Pneumococcal Serotypes Contained in V116
Description: The percentage of participants with ≥4-fold rise from baseline to post-vaccination with V116 and PCV15+PPSV23 in serotype-specific OPA responses for pneumococcal serotypes contained in V116 was calculated using MOPA. The 13 common pneumococcal serotypes in both V116 and PCV15 + PPSV23 were as follows: 3, 6A, 7F, 8, 9N, 10A, 11A, 12F, 17F, 19A, 20A, 22F, and 33F. The 8 unique pneumococcal serotypes in V116 were as follows: 15A, 15C, 16F, 23A, 23B, 24F, 31, and 35B.
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V116 + Placebo | PCV15 + PPSV23
Number analyzed (Participants) | 386 | 130
Percentage of Participants
  Serotype 3: number analyzed (Participants) | 334 | 102
  Serotype 3 | 70.1 [64.8 to 74.9] | 63.7 [53.6 to 73.0]
  Serotype 6A: number analyzed (Participants) | 297 | 82
  Serotype 6A | 79.1 [74.1 to 83.6] | 79.3 [68.9 to 87.4]
  Serotype 7F: number analyzed (Participants) | 341 | 107
  Serotype 7F | 78.3 [73.5 to 82.6] | 63.6 [53.7 to 72.6]
  Serotype 8: number analyzed (Participants) | 344 | 103
  Serotype 8 | 84.6 [80.3 to 88.2] | 82.5 [73.8 to 89.3]
  Serotype 9N: number analyzed (Participants) | 336 | 107
  Serotype 9N | 74.7 [69.7 to 79.3] | 58.9 [49.0 to 68.3]
  Serotype 10A: number analyzed (Participants) | 327 | 98
  Serotype 10A | 74.9 [69.9 to 79.5] | 70.4 [60.3 to 79.2]
  Serotype 11A: number analyzed (Participants) | 326 | 100
  Serotype 11A | 76.7 [71.7 to 81.2] | 49.0 [38.9 to 59.2]
  Serotype 12F: number analyzed (Participants) | 343 | 107
  Serotype 12F | 94.2 [91.1 to 96.4] | 85.0 [76.9 to 91.2]
  Serotype 17F: number analyzed (Participants) | 327 | 101
  Serotype 17F | 89.6 [85.8 to 92.7] | 76.2 [66.7 to 84.1]
  Serotype 19A: number analyzed (Participants) | 337 | 102
  Serotype 19A | 68.0 [62.7 to 72.9] | 68.6 [58.7 to 77.5]
  Serotype 20A: number analyzed (Participants) | 335 | 97
  Serotype 20A | 66.9 [61.5 to 71.9] | 42.3 [32.3 to 52.7]
  Serotype 22F: number analyzed (Participants) | 322 | 102
  Serotype 22F | 74.8 [69.7 to 79.5] | 57.8 [47.7 to 67.6]
  Serotype 33F: number analyzed (Participants) | 330 | 100
  Serotype 33F | 78.5 [73.7 to 82.8] | 58.0 [47.7 to 67.8]
  Serotype 15A: number analyzed (Participants) | 309 | 95
  Serotype 15A | 67.6 [62.1 to 72.8] | 29.5 [20.6 to 39.7]
  Serotype 15C: number analyzed (Participants) | 335 | 105
  Serotype 15C | 86.0 [81.8 to 89.5] | 72.4 [62.8 to 80.7]
  Serotype 16F: number analyzed (Participants) | 334 | 96
  Serotype 16F | 65.6 [60.2 to 70.7] | 16.7 [9.8 to 25.6]
  Serotype 23A: number analyzed (Participants) | 261 | 76
  Serotype 23A | 71.3 [65.4 to 76.7] | 52.6 [40.8 to 64.2]
  Serotype 23B: number analyzed (Participants) | 341 | 106
  Serotype 23B | 87.7 [83.7 to 91.0] | 49.1 [39.2 to 59.0]
  Serotype 24F: number analyzed (Participants) | 293 | 81
  Serotype 24F | 41.6 [35.9 to 47.5] | 6.2 [2.0 to 13.8]
  Serotype 31: number analyzed (Participants) | 344 | 99
  Serotype 31 | 77.0 [72.2 to 81.4] | 16.2 [9.5 to 24.9]
  Serotype 35B: number analyzed (Participants) | 337 | 102
  Serotype 35B | 64.4 [59.0 to 69.5] | 5.9 [2.2 to 12.4]

9. Secondary Outcome: Percentage of Participants With ≥4-fold Change From Baseline to Post-Vaccination With V116 and PCV15 + PPSV23 in Serotype Specific IgG Responses for Pneumococcal Serotypes Contained in V116
Description: The percentage of participants with ≥4-fold rise from baseline to post-vaccination with V116 and PCV15+PPSV23 in serotype-specific OPA responses for pneumococcal serotypes contained in V116 was calculated using Pn ECL assay. The 13 common pneumococcal serotypes in both V116 and PCV15 + PPSV23 were as follows: 3, 6A, 7F, 8, 9N, 10A, 11A, 12F, 17F, 19A, 20A, 22F, and 33F. The 8 unique pneumococcal serotypes in V116 were as follows: 15A, 15C, 16F, 23A, 23B, 24F, 31, and 35B.
Time Frame: as for outcome 6
Population: The population analyzed was all randomized participants without deviations from the protocol that may substantially affect the results of the immunogenicity endpoints. Deviations include, but are not limited to the following: failure to receive the study vaccine, receiving incorrect clinical material per the randomization schedule, or taking prohibited medications or vaccines prior to vaccination or blood sample collection outside the designated window.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V116 + Placebo | PCV15 + PPSV23
Number analyzed (Participants) | 386 | 130
Percentage of Participants
  Serotype 3: number analyzed (Participants) | 365 | 111
  Serotype 3 | 57.8 [52.6 to 62.9] | 54.1 [44.3 to 63.6]
  Serotype 6A: number analyzed (Participants) | 366 | 111
  Serotype 6A | 81.1 [76.8 to 85.0] | 86.5 [78.7 to 92.2]
  Serotype 7F: number analyzed (Participants) | 366 | 111
  Serotype 7F | 88.8 [85.1 to 91.8] | 83.8 [75.6 to 90.1]
  Serotype 8: number analyzed (Participants) | 366 | 111
  Serotype 8 | 82.2 [77.9 to 86.0] | 83.8 [75.6 to 90.1]
  Serotype 9N: number analyzed (Participants) | 366 | 111
  Serotype 9N | 86.9 [83.0 to 90.2] | 78.4 [69.6 to 85.6]
  Serotype 10A: number analyzed (Participants) | 366 | 111
  Serotype 10A | 86.3 [82.4 to 89.7] | 79.3 [70.5 to 86.4]
  Serotype 11A: number analyzed (Participants) | 366 | 111
  Serotype 11A | 79.8 [75.3 to 83.8] | 63.1 [53.4 to 72.0]
  Serotype 12F: number analyzed (Participants) | 366 | 111
  Serotype 12F | 82.8 [78.5 to 86.5] | 69.4 [59.9 to 77.8]
  Serotype 17F: number analyzed (Participants) | 366 | 111
  Serotype 17F | 93.2 [90.1 to 95.5] | 82.9 [74.6 to 89.4]
  Serotype 19A: number analyzed (Participants) | 366 | 111
  Serotype 19A | 64.2 [59.1 to 69.1] | 73.0 [63.7 to 81.0]
  Serotype 20A: number analyzed (Participants) | 366 | 111
  Serotype 20A | 83.1 [78.8 to 86.8] | 75.7 [66.6 to 83.3]
  Serotype 22F: number analyzed (Participants) | 366 | 111
  Serotype 22F | 85.0 [80.9 to 88.5] | 83.8 [75.6 to 90.1]
  Serotype 33F: number analyzed (Participants) | 366 | 111
  Serotype 33F | 87.2 [83.3 to 90.4] | 79.3 [70.5 to 86.4]
  Serotype 15A: number analyzed (Participants) | 366 | 111
  Serotype 15A | 88.3 [84.5 to 91.4] | 44.1 [34.7 to 53.9]
  Serotype 15C: number analyzed (Participants) | 366 | 110
  Serotype 15C | 88.5 [84.8 to 91.6] | 75.5 [66.3 to 83.2]
  Serotype 16F: number analyzed (Participants) | 366 | 110
  Serotype 16F | 85.8 [81.8 to 89.2] | 7.3 [3.2 to 13.8]
  Serotype 23A: number analyzed (Participants) | 366 | 111
  Serotype 23A | 88.3 [84.5 to 91.4] | 37.8 [28.8 to 47.5]
  Serotype 23B: number analyzed (Participants) | 366 | 111
  Serotype 23B | 81.7 [77.3 to 85.5] | 43.2 [33.9 to 53.0]
  Serotype 24F: number analyzed (Participants) | 366 | 111
  Serotype 24F | 82.0 [77.6 to 85.8] | 2.7 [0.6 to 7.7]
  Serotype 31: number analyzed (Participants) | 366 | 111
  Serotype 31 | 83.1 [78.8 to 86.8] | 9.9 [5.1 to 17.0]
  Serotype 35B: number analyzed (Participants) | 366 | 111
  Serotype 35B | 79.5 [75.0 to 83.5] | 0.9 [0.0 to 4.9]

ADVERSE EVENTS:
Time Frame: Up to ~ 194 Days following Visit 2 (Day 1)
Description: The all-cause mortality population includes all randomized participants. The SAE and AE analysis population includes all participants who were randomized and received at least 1 dose of study intervention.
Arm/Group | V116 + Placebo | PCV15 + PPSV23
All-Cause Mortality (participants affected / at risk) | 0/387 | 0/131
Serious Adverse Events (participants affected / at risk) | 10/386 | 7/130
Other Adverse Events (participants affected / at risk) | 240/386 | 112/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V116 + Placebo (N=386) | PCV15 + PPSV23 (N=130)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V116 + Placebo (N=386) | PCV15 + PPSV23 (N=130)
Fatigue (General disorders) | 118 (152) | 59 (75)
Injection site erythema (General disorders) | 39 (41) | 33 (36)
Injection site pain (General disorders) | 200 (223) | 102 (176)
Injection site swelling (General disorders) | 33 (37) | 46 (55)
Myalgia (Musculoskeletal and connective tissue disorders) | 42 (50) | 20 (22)
Headache (Nervous system disorders) | 94 (116) | 36 (46)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/80/NCT05696080/Prot_SAP_000.pdf